CLINICAL TRIAL: NCT01009879
Title: Human TNFa-Induced Pre-B Cell Bone Marrow Emigrants
Brief Title: Human Tumor Necrosis Factor Alpha (TNFa)-Induced Pre-B Cell Bone Marrow Emigrants
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects were enrolled
Sponsor: University of Pittsburgh (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, MarcLevesque, Associate Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AMGEN 2006_1112
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; B lymphocytes
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg SQ qweek
  Other Names: ENBREL

SUMMARY:
The purpose of the study is to determine the effects of TNF (tumor necrosis factor; a mediator of inflammation) on B cells in patients with rheumatoid arthritis. TNF and B cells are important in rheumatoid arthritis because they both appear to be involved in causing rheumatoid arthritis.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of the study is to identify early B cell bone marrow emigrants in the peripheral blood of adults with rheumatoid arthritis (RA) receiving etanercept.

Hypotheses: We believe that the peripheral blood of RA patients contain early B cell bone marrow emigrants. We believe that these early B cell bone marrow emigrants are induced by TNFα.

Primary Endpoint: The primary endpoint of the study is quantification of CD34+/CD19+ early B cell bone marrow emigrants in the peripheral blood of subjects.

Study Design: Open-label, One Arm, Phase IV study of 12 RA patients with active disease receiving etanercept.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA) patients will be eligible for the study if they meet ACR criteria for a diagnosis of RA (Arnett et al. 1988. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis & Rheumatism 31:315.) and have active disease (≥ 6 tender and/or swollen joints).
* Subjects must be ≥ 18 years of age.
* Subjects must be rheumatoid factor (RF) positive (any RF titer greater than the upper limits of normal) and/or anti-CCP antibody positive (any anti-CCP titer greater than the upper limits of normal). Subjects must have a negative TB skin test at entry into the study or a negative screening chest x-ray if the PPD test is inconclusive (borderline, reactive but non-diagnostic) or in prior BCG inoculated subjects. Female subjects of child bearing potential (excludes those that are surgically sterile or at least 5 years postmenopausal) must have a negative pregnancy test (serum β-HCG). Sexually active subjects of childbearing potential must agree to use medically acceptable forms of contraception during screening and throughout the study.
* Subjects or a designee must have the ability to self-inject ENBREL or a care-giver at home who can administer subcutaneous injections. Subjects must be willing to remain on ENBREL (50 mg SQ qweek) for at least 12 weeks and have not taken anti-rheumatic agents (DMARDS and/or corticosteroids) besides NSAIDs for the previous 4 weeks.
* The subject must be able and willing to give written informed consent and comply with the requirements of the study protocol and must authorize release and use of protected health information. Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* RA patients will be excluded if they have a history of congestive heart failure, recurrent or active infection, a positive PPD, history of neurologic disease, Felty's syndrome, hematologic malignancy or liver disease.
* RA patients will be excluded if they have a WBC count < 4.0, Hct < 30 or liver profile abnormalities (> 2x normal values of AST, ALT, TBili and/or APhos).
* RA patients will be excluded if they have been previously treated with anti-TNFα therapy (ENBREL, infliximab or adalimumab), IL-1ra, abatacept or B and T cell depleting therapies including rituximab or alemtuzumab. Subjects who have previously received other DMARD therapies including methotrexate, leflunomide, sulfasalazine, hydroxychloroquine, gold, penicillamine, cyclosporine A, and cyclophosphamide must not have taken one of these medications within the past 30 days prior to instituting ENBREL.
* General: Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit. Subjects who have known hypersensitivity to Enbrel or any of its components or who is known to have antibodies to etanercept.

Prior or concurrent cyclophosphamide therapy. Concurrent sulfasalazine therapy. Known HIV-positive, mycobacterial disease, active severe infections, untreated Lyme disease, severe comorbidities, history of TB or TB exposure, chronic hepatitis B or hepatitis C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy, history of recent alcohol or substance abuse (< 1 year), pregnant or lactating females and/or use of a live vaccine 90 days prior to, or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to quantify early B cell bone marrow emigrants in the peripheral blood of adults with rheumatoid arthritis (RA) before and after etanercept therapy. | 12 weeks

SECONDARY OUTCOMES:
Secondary objectives will include granulocyte numbers, serum cytokine (CRP, IL-1β and TNFα) levels, rheumatoid arthritis disease activity and changes in anti-CCP and RF levels before and after etanercept therapy. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc C Levesque, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh - Oakland Falk Clinic, Pittsburgh, Pennsylvania, United States